CLINICAL TRIAL: NCT07248683
Title: Application of Ultrasound-Guided Midline Combined With Spaced Retrieval Training in Radial Artery Puncture and Catheterization for Standardized-Trained Residents：A Randomized Sequential Allocation Study
Brief Title: Application of Intermittent Training in Radial Artery Puncture and Catheterization Skills Under Ultrasound-Guided Line Guidance
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: General Hospital of Ningxia Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Haoyao Ren--2025-11
Record Dates: First submitted 2025-11-18; First posted 2025-11-25 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-08

CONDITIONS: Learning and Memorization of Radial Artery Puncture and Catheterization Guided by Ultrasound Midline

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interval Training Group (Experimental): All participants underwent centralized training. The intermittent retraining group performed fixed-interval repeated training, executing the same tasks daily on days 3, 7, and 14.
  Interventions: Other: Intermittent Retraining
- Non-interval retraining (Experimental): Through centralized training, it was confirmed that all trainees had mastered the steps of radial artery puncture and catheterization guided by the midline ultrasound. A test validated the students' proficiency in this procedure. The non-intermittent retraining group will not undergo intermittent training during the following week.
  Interventions: Other: Non-interval retraining

INTERVENTIONS:
Other: Intermittent Retraining — Through basic skills training and testing, it was confirmed that all trainees had mastered the procedural steps for radial artery puncture and catheterization guided by ultrasound midline imaging. Testing also validated the students' proficiency in performing this procedure. The intermittent retraining group underwent repeated training at fixed intervals, performing the same tasks daily on days 3, 7, and 14.
  Arms: Interval Training Group
Other: Non-interval retraining — Through basic skills training and testing, it was confirmed that all trainees had mastered the procedural steps for radial artery puncture and catheterization guided by ultrasound midline imaging. Testing also validated the students' proficiency in performing this procedure. The non-intermittent retraining group did not repeat the same tasks.
  Arms: Non-interval retraining

SUMMARY:
This study aims to investigate medical students' mastery of radial artery puncture and catheterization skills guided by the midline on ultrasound when using scenario simulation combined with intermittent training, and to compare this approach with traditional teaching methods.

DETAILED DESCRIPTION:
With the continuous advancement of modern anesthesiology and critical care medicine, arterial monitoring has become an integral part of clinical anesthesia management. During anesthesia, functions such as arterial blood pressure monitoring and arterial blood gas analysis enable real-time surveillance of vital signs, playing a crucial role particularly in the anesthesia management and postoperative monitoring of high-risk patients. The radial artery, being a superficial and easily accessible vessel, has become one of the commonly used arterial puncture sites in clinical practice. Furthermore, this technique is a mandatory skill for residents in standardized training programs within anesthesiology departments. However, as an invasive procedure, it demands high proficiency from the operator and carries significant risks of complications such as infection, hematoma, thrombosis, and arterial spasm. Radial artery catheterization poses a challenge for residents, making it essential to establish a straightforward and clear teaching strategy.The success rate of ultrasound-guided radial artery puncture is influenced by operator experience, particularly among resident physicians. Although ultrasound with a "midline" feature can assist in puncture, catheter placement remains challenging, and the effectiveness of their mastery requires further study. Current training programs exhibit gaps, with clinical settings predominantly relying on intensive learning sessions that yield poor skill retention. Interval learning, despite its advantages, is underutilized. Given the clinical workload constraints of residents, sustained practice after intensive training is challenging. Therefore, designing and implementing an intermittent training program for ultrasound-guided radial artery catheterization is highly significant. This approach aims to combine the strengths of both intensive and intermittent training to enhance residents' skills, reduce complications, ensure patient safety, and provide departments with a new, effective training method.

ELIGIBILITY:
Inclusion and Exclusion Criteria for Study Participants (Resident Trainees) I. Inclusion Criteria Identity and Qualifications: Resident physicians undergoing standardized training in this department.

Training Stage: Resident physicians who have not yet independently performed ultrasound-guided radial artery puncture and catheterization procedures.

Willingness to Learn: Voluntary participation in this "Ultrasound-Guided Radial Artery Catheterization" training program with full understanding of the research content.

Informed Consent: Have signed a written informed consent form agreeing to participate in this study and comply with protocol requirements.

Basic Requirements: Possess good hand-eye coordination and learning ability, capable of cooperating to complete the entire training course and data collection.

II. Exclusion Criteria Prior Experience: Residents who have previously independently completed more than 5 cases or have systematically studied ultrasound-guided radial artery puncture and catheterization techniques.

Skill Level: Residents who achieved a high pre-test performance score or demonstrated consistent success in performing ultrasound-guided radial artery catheterization prior to the study.

Cognitive or Motor Impairment: Residents with severe cognitive dysfunction, motor impairment, or a history of psychiatric disorders that may compromise training efficacy assessment.

Time Commitment and Compliance: Individuals unable to guarantee completion of the prescribed training program, practical exercises, and follow-up evaluations.

Other Conditions: Participants deemed unsuitable for this study by the investigator due to other reasons (e.g., rotation schedule conflicts, inability to coordinate personal time, etc.).

Inclusion and Exclusion Criteria for Study Subjects (Patients Undergoing Radial Artery Catheterization)

I. Inclusion Criteria

Age: Generally ≥18 years old. Clinical Indications: Patients requiring invasive arterial pressure monitoring via radial artery puncture and catheterization due to surgical procedures, critical condition monitoring, or blood gas analysis.

Vascular Criteria: Palpable radial artery pulse on the puncture side, negative modified Allen test (or adequate ulnar artery compensation as determined by current guidelines).

Informed Consent: Patient or authorized family member fully understands the study purpose and procedures, and has signed a written informed consent form.

Cooperation Capacity: Able to cooperate throughout the radial artery puncture and catheterization procedure.

II. Exclusion Criteria Contraindications for Puncture: History of thrombosis, aneurysm, or arteriovenous fistula at the puncture site; skin infection, laceration, burn, or severe scar tissue at the puncture site.

Circulatory Impairment: Severe shock, hypovolemic state, or anticipated difficulty with radial artery puncture.

Coagulation Abnormalities: Significant bleeding tendency, marked thrombocytopenia, or ongoing anticoagulant/antiplatelet therapy without discontinuation.

Abnormal vascular anatomy: Preliminary ultrasound assessment indicates severe tortuosity, malformation, excessively narrow diameter, or other significant anatomical variations in the radial artery that may compromise puncture success or safety.

Special circumstances: Requirement for simultaneous bilateral radial artery catheterization; or other situations deemed unsuitable for this teaching procedure by the investigator.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-11-20 (Estimated); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
First Attempt Catheterization Success Rate | The fourteenth day after the unified training
  The percentage of cases where the operator successfully punctures the target vessel (specifically the radial artery in my study) on the first attempt and advances the catheter to the desired position. This process requires no additional puncture attempts, catheter adjustments, or encounters procedural failure (such as unsuccessful vessel entry, guidewire/catheter entanglement, abnormal positioning, or immediate complications like hematoma formation).
First-Attempt Radial Artery Catheterization Success Rate | The 14th day after training
  First-Attempt Success Rate of Radial Artery Catheterization Guided by Ultrasound Median Line
Incidence of complications | The 14th day after training
  Incidence of Complications in Radial Artery Puncture and Catheterization Guided by Ultrasound Midline